CLINICAL TRIAL: NCT06808373
Title: The Effect of Hypnosis on Healing in Patients Undergoing Phase I Periodontal Therapy
Brief Title: The Effect of Hypnosis on Periodontal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Kübra Karaçam, assist. prof., Afyonkarahisar Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBUSAH-GETAT 2024-054
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Peridontal Disease; Dental Anxiety
Keywords: periodontitis, hypnosis, dental anxiety
MeSH Terms: conditions — Periodontitis | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hypnosis (Experimental): Hypnosis will be applied to patients with periodontitis.
  Interventions: Behavioral: hypnosis

INTERVENTIONS:
Behavioral: hypnosis — Hypnosis will be applied to periodontitis patients

SUMMARY:
Treatment of periodontal diseases relies on the mechanical removal of microbial dental plaque, calculus, and necrotic cementum from root surfaces in both supra- and subgingival areas to control inflammation in periodontal tissues. As in all dental treatments, dental phobia and dental anxiety are common challenges in initial periodontal therapy. Hypnosis is among the traditional non-pharmacological behavior management techniques used to manage stress and improve pain tolerance. It is known that hypnosis is effective in anxiety control in dentistry. The use of salivary levels of inflammatory mediators released during the disease is a valid method for assessing the progression of periodontal disease and healing after treatment. In this study, the effect of hypnosis on healing in patients undergoing Phase I periodontal therapy will be evaluated by comparing the mean differences in cytokine levels between case and control groups

ELIGIBILITY:
Inclusion Criteria:

Being between the ages of 20-65 Not having any systemic disease Having chronic periodontal disease Having the ability to understand the study and answer questions

Exclusion Criteria:

Having any systemic disease Being under 20 or over 65 Not having any periodontal disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
measurement of cytokine levels | Pre-treatment (day 0), post-treatment (day 0) and 8 weeks post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University Faculty of Dentistry, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No